CLINICAL TRIAL: NCT02918682
Title: The Effects of a Multi-component Intervention on the Functional Capacity, Upper and Lower-body Muscle Strength, Balance and Gait in Frail Community-dwelling Older People: a Randomized Clinical Trial
Brief Title: A Multi-component Intervention in Frail Community-dwelling Older People
Acronym: MIF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Prof Daniela Cristina Carvalho de Abreu, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 932.043
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Frail Elderly; Exercise Therapy; Physical Therapy Techniques

STUDY DESIGN:
Intervention Model Description: the participants do not need to perform the first phase or can advance to the second phase if they have obtained the following results in the balance and functional tests: 1. Gait speed of 0.8 m/s and walking 30 meters without stopping; 2. Ability to perform the stand up and sit down test from the chair five times properly within less than 15 seconds; 3. Maintaining the FFEO stance for 30 seconds and the Tandem EO stance for more than 5 seconds; 4. Having sitting stability limits with eyes open; 5. In upright position, able to bend the trunk forward, standing parallel to a wall, between 16.5 - 32 cm but stable. For the muscle strength: being able to perform hip flexion with 50% of 1 repetition maximum (RM) for 8 repetitions; hip extension with 50% of 1RM for 8 repetitions; hip abduction without load but at least for 8 repetitions; knee extension with 50% of 1RM for 8 repetitions; knee flexion with 50 % of 1RM for 8 repetitions;
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The multimodal intervention protocol is described separated by day (1 to 24) and by weeks (1 to 12). Each session was built to last between 50 and 60 minutes.
  Interventions: Other: Exercise - FIRST PHASE; Other: Exercise - SECOND PHASE; Other: Exercise - FOURTH PHASE; Other: Exercise - THIRD PHASE
- Control Group (No Intervention): Participants from the control group will not perform any kind of physical exercise.

INTERVENTIONS:
Other: Exercise - FIRST PHASE — the participants do not need to perform the first phase or can advance to the second phase if they have obtained the following results in the balance and functional tests: 1. Gait speed of 0.8 m/s and walking 30 meters without stopping; 2. Ability to perform the stand up and sit down test from the chair five times properly within less than 15 seconds; 3. Maintaining the FFEO stance for 30 seconds and the Tandem EO stance for more than 5 seconds; 4. Having sitting stability limits with eyes open; 5. In upright position, able to bend the trunk forward, standing parallel to a wall, between 16.5 - 32 cm but stable. For the muscle strength: being able to perform hip flexion with 50% of 1 repetition maximum (RM) for 8 repetitions; hip extension with 50% of 1RM for 8 repetitions; hip abduction without load but at least for 8 repetitions; knee extension with 50% of 1RM for 8 repetitions; knee flexion with 50 % of 1RM for 8 repetitions;
  Arms: Exercise Group
Other: Exercise - SECOND PHASE — the participants do not need to perform the second phase or can advance to the third phase if they have obtained the following results in the balance and functional tests: 1. Gait speed of 0.8-1 m/s and ability to walk 60 meters; 2. Ability to perform the stand up and sit down test from the chair five times properly within less than 15 seconds; 3. Maintaining the FFEO and FFEC stance for more than 5 seconds and the Tandem EO stance for 10-20 seconds; 4. Having sitting stability limits with eyes closed; 5. Being able to bend the trunk forward, standing parallel to a wall, between 20-32 cm ad being stable. For muscle strength: being able to perform hip flexion with 60% of 1 RM for 8 repetitions; hip extension with 60% of 1RM for 8 repetitions; hip abduction without load but between 8-12 repetitions; knee extension with 60% of 1RM for 8 repetitions; knee flexion with 60% of 1RM for 8 repetitions;
  Arms: Exercise Group
Other: Exercise - FOURTH PHASE — at the end of the exercise protocol, the participants who have reached the fourth phase must be able to achieve: 1. Gait speed of 0.8-1 m/s and able to walk 90 meters; 2. Stand up and sit down five times from the chair properly within less than 15 seconds; 3. TUG performance less than 14 seconds; 4. Maintenance of 30 seconds in FFEO and FFEC stance, maintenance of 30 seconds in Tandem EO and Tandem EC stance, maintenance of the single-leg stance for more than 21 seconds; 5. Normal sitting stability limits with eyes closed; 6. Bending the trunk forward, standing parallel to a wall, more than 32 cm and being stable. For muscle strength: able to perform hip flexion with 70% of 1 RM for 6-10 repetitions; hip extension with 70% of 1RM for 6-10 repetitions; hip abduction with 40-60% of 1RM for 8-12 repetitions; knee extension with 70% of 1RM for 6-10 repetitions; knee flexion with 70% of 1RM for 6-10 repetitions.
  Arms: Exercise Group
Other: Exercise - THIRD PHASE — participants do not need to perform the third phase or can advance to the fourth phase if they have obtained: 1 Gait speed of 0.8-1 m/s and walk 90 meters; 2 perform the stand up and sit down five times from the chair properly within less than 15 seconds; 3 Performing the TUG test within less than 14 seconds; 4 Maintaining the FFEO and FFEC stance for 30 seconds, maintaining the Tandem EO and Tandem EC stance for 30 seconds and maintaining the single-leg stance for more than 20 seconds; 5 Having sitting stability limits with eyes closed; 6 In the upright position, to bend the trunk forward, standing parallel to a wall, more than 32 cm and being stable. For the muscle strength test, perform hip flexion with 60 % of 1 RM for 8-12 repetitions; hip extension with 60 % of 1RM for 8-12 repetitions; hip abduction without load or 5% of 1RM for hip abductor and between 8-12 repetitions; knee extension with 60 % of 1RM for 8-12 repetitions; knee flexion with 60 % of 1RM for 8-12 repetitions;
  Arms: Exercise Group

SUMMARY:
This study evaluates if a multi-component intervention, respecting the characteristics of frail older person and increasing intensity and challenge of exercises according to frail older person capacity/evolution will induce better functional results than a multi-component intervention specific to lower body. the volunteers will be randomized into experimental group and control group.

DETAILED DESCRIPTION:
The interventions are separated by day (1 to 24) and by weeks (1 to 12). Each session was built to last between 50 and 60 minutes, beginning with a warming up. In the table are described the exercise as well as the support necessary to perform the exercise safely and necessary equipment (accessories). In cases where a minimum load is required the same are also described in the multimodal intervention protocol (load).

In relation to strength training in the multimodal intervention protocol is described how the progression of intensity will be held. Additional to the load progression suggested, the 1 maximal repetition test will be applied every 4 weeks for adjustment of the loads according to strength gain from each volunteer.

The suggested protocol is based on balance exercises and strength but, in a careful manner, were included functional and mobilization exercises to ensure greater diversity.

Multimodal intervention protocol:

1. a week

   Day 1. Balance Training 1.1 P: Seated on the chair; E: Position Adjustments, (Anterior-posterior, medial-lateral); S: Yes (parallel bar) 1.2 P: Seated on the chair; E: Hip mobilization, Anterior- posterior; S: Yes(parallel bar)

   Strength Training 1.1 P: Dorsal Decubitus; E: Hip Flexion 1.2 P:Lateral Decubitus; E: Hip Abduction 1.3 P:Seated on the chair; E: Knee Extension 1.4 P:Seated on the chair; E: Dorsiflexion/ Plantar Flexion 1.5 P:Seated on the chair; E: Trunk stabilization; A: Stick
2. sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 2. Balance Training 2.1 P: Seated on the chair; E: Position Adjustments (Anterior-posterior, medial-lateral);S: Yes(parallel bar) 2.2 P: Seated on the chair; E: Hip mobilization Anterior- posterior; S: Yes(parallel bar)

Strength Training 2.1 P: Ventral Decubitus; E: Hip Extension (hollowing) 2.2 P:Lateral Decubitus; E: Hip Aduction 2.3 P: Standing; E: Semi-squat; A: peanut ball 2.4 P: Standing; E: Knee Flexion; S: Yes (parallel bar or back rest)

2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

2a week

Day 3. Balance Training 3.1 P:Seated on the chair; E: Trunk mobilization Latero-lateral; S: Yes (parallel bar) 3.2 P:Seated on the chair; E: Trunk mobilization Anterior-posterior; S: Yes(parallel bar) 3.3 P: Standing; E:Romberg- feet together, semi-tandem, tandem; S: Yes(parallel bar) Strength Training 3.1 P: Dorsal Decubitus; E: Hip Flexion 3.2 P:Lateral Decubitus; E: Hip Abduction 3.3 P:Seated on the chair; E: Knee Extension 3.4 P:Seated on the chair; E: Dorsiflexion/ Plantar Flexion 3.5 P:Seated on the chair; E: Trunk stabilization; A: Stick 2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 4. Balance Training 4.1 P:Seated on the chair; E: Trunk mobilization Latero-lateral; S: Yes (parallel bar) 4.2 P:Seated on the chair; E: Trunk mobilization Anterior-posterior; S: No 4.3 P: Standing; E:Romberg- feet together, semi-tandem, tandem; S: Yes(parallel bar) Strength Training 4.1 P:Ventral Decubitus; E: Hip Extension (hollowing) 4.2 P:Lateral Decubitus; E: Hip Aduction 4.3 P: Standing; E: Semi-squat; A: peanut ball 4.4 P: Standing; E: Knee Flexion; S: Yes (parallel bar or back rest )

2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

3a week

Day 5. Balance Training 5.1 P: Standing; E: Side step walking; S: Yes (parallel bar) 5.2 P: Standing; E: Sitting to standing; S: Yes (parallel bar or) back rest 5.3 P: Standing; E:Romberg- feet together, semi-tandem, tandem; S: No 5.4 P: Table pose (Time: 60s )

Strength Training 5.1 P: Dorsal Decubitus; E: Hip Flexion 5.2 P:Lateral Decubitus; E: Hip Abduction 5.3 P:Seated in the chair; E: Knee Extension 5.4 P:Seated on the chair; E: Dorsiflexion/ Plantar Flexion

2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 6. Balance Training 6.1 P: Standing; E:Side step walking; S: Yes (parallel bar) 6.2 P: Standing; E: Sitting to standing; S: Yes (parallel bar or back rest) 6.3 P: Standing; E:Romberg- feet together, semi-tandem, tandem; S: No 6.4 P: Table pose(Time: 60s )

Strength Training 6.1 P:Ventral Decubitus; E: Hip Extension (hollowing + one leg up) 6.2 P:Lateral Decubitus; E: Hip Aduction 6.3 P: Standing; E: Semi-squat; A: peanut ball 6.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest)

2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

4a week

Day 7. Balance Training 7.1 P: Standing; E: Walk to Front and Back; S: Yes (parallel bar) 7.2 P: Standing; E: Side step walking; S: No 7.3 P: Seated on the chair; E: Sit to standing; S: Standing: No; Sitting: Yes (parallel bar or back rest) 7.4 P: Table pose(Time: 60s ) 7.5 P: Standing; E:Romberg- feet together, semi-tandem, tandem; S: No

Strength Training 7.1 P: Dorsal Decubitus; E: Hip Flexion 7.2 P:Lateral Decubitus; E: Hip Abduction 7.3 P:Seated in the chair; E: Knee Extension 7.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes(parallel bar or back rest )

2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 8. Balance Training 8.1 P: Standing; E: Walk to Front and Back; S: Yes (parallel bar) 8.2 P: Standing; E: Side step walking; S: No 8.3 P: Seated on the chair; E: Sit to standing; S: Standing: No; Sitting: Yes(parallel bar or back rest) 8.4 P: Table pose(Time: 60s ) 8.5 P: Standing; E:Romberg- feet together, semi-tandem, tandem; S: No

Strength Training 8.1 P:Ventral Decubitus; E: Hip Extension (hollowing + one leg up) 8.2 P:Lateral Decubitus; E: Hip Aduction 8.3 P: Standing; E: Semi-squat; L: 0.5 Kg 8.4 P: Standing; E: Knee Flexion; S: No

2 sets, 12 repetitions, 50% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

5a week

Day 9. Balance Training 9.1 P: Seated on the chair; E: Sitting to standing; S: No 9.2 P: Standing; E: One leg stance; S: Yes(parallel bar) 9.3 P: Standing; E: Walk to Front and Back; S: No 9.4 P: Standing; E: Tandem position; S: No + ocular fixation

Strength Training 9.1 P: Dorsal Decubitus; E:Hip Flexion 9.2 P:Lateral Decubitus; E: Hip Abduction 9.3 P:Seated on the chair; E: Knee Extension 9.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes (parallel bar or back rest)

3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 10. Balance Training 10.1 P: Seated on the chair; E: Sitting to standing; S: No 10.2 P: Standing; E: One leg stance; S: Yes (parallel bar) 10.3 P: Standing; E: Walk to Front and Back; S: No 10.4 P: Standing; E: Tandem position; S: No + ocular fixation

Strength Training 10.1 P: Ventral Decubitus; E: Hip Extension (Table position) 10.2 P:Lateral Decubitus; E: Hip Aduction 10.3 P:Standing; E: Semi-squat; S:No; L:1 Kg 10.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest)

3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

6a week

Day 11. Balance Training 11.1 P: Standing; E:Crossed Gait (Braiding); S:Yes (parallel bar) 11.2 P: Standing; E: Turn 90º or 180º; S:Yes(parallel bar) 11.3 P: Standing; Reactive Balance (Ankle, Hip, Step); S:Yes(parallel bar) 11.4 P:Standing; E:Romberg- feet together; S: No+ eyes closed 11.5 P: Standing; E: One leg stance; S: No

Strength Training 11.1 P: Dorsal Decubitus; E:Hip Flexion 11.2 P:Lateral Decubitus; E: Hip Abduction 11.3 P:Seated on the chair; E: Knee Extension 11.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes(parallel bar or back rest)

3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 12. Balance Training 12.1 P: Standing; E:Crossed Gait (Braiding); S:Yes (parallel bar) 12.2 P: Standing; E: Turn 90º or 180º; S:Yes(parallel bar) 12.3 P: Standing; Reactive Balance (Ankle, Hip, Step); S:Yes(parallel bar) 12.4 P:Standing; E:Romberg- feet together; S: No+ eyes closed 12.5 P: Standing; E: One leg stance; S: No

Strength Training 12.1 P: Ventral Decubitus; E: Hip Extension (Table position) 12.2 P:Lateral Decubitus; E: Hip Aduction 12.3 P:Standing; E: Semi-squat; S:No; L:1 Kg 12.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest) 3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

7a week

Day 13. Balance Training 13.1 P: Standing; E:Walk with Hip flexion 90o like soldier); S: Yes, (parallel bar) 13.2 P: Standing; E: Turn 180º ou 360º; S:Yes(parallel bar) 13.3 P: Standing; E:Walk (6 meters) increasing step length; S: No 13.4 P: Standing; E:Tandem Posture; S: No 13.5 P: Standing; E: One leg stance; S: No + eyes closed

Strength Training 13.1 P: Dorsal Decubitus; E: Hip Flexion 13.2 P:Lateral Decubitus; E: Hip Abduction 13.3 P:Seated on the chair; E: Knee Extension 13.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes(parallel bar or back rest)

3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 14. Balance Training 14.1 P: Standing; E:Walk with Hip flexion 90o like soldier); S:Yes(parallel bar) 14.2 P: Standing; E: Turn 180º ou 360º; S:Ye(parallel bar)s 14.3 P: Standing; E:Walk (6 meters) increasing step length; S: No 14.4 P: Standing; E:Tandem Posture; S: No 14.5 P: Standing; E: One leg stance; S: No + eyes closed

Strength Training 14.1 P: Ventral Decubitus; E: Hip Extension (Table position) 14.2 P:Lateral Decubitus; E: Hip Aduction 14.3 P:Standing; E: Semi-squat; S:No; L:1 Kg 14.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest)

3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

8a week

Day 15. Balance Training 15.1 P: Standing; E:Walk with Hip flexion 90o like soldier); S:No 15.2 P: Standing; E: Tandem Gait; S: Yes(parallel bar) 15.3 P: Standing; E: Step up and down; S: No 15.4 P: Seated on the chair; E:TUG habitual walk speed; S: No 15.5 P:Standing; E:Romberg- feet together; S: No+ ball reach

Strength Training 15.1 P: Dorsal Decubitus; E: Hip Flexion 15.2 P:Lateral Decubitus; E: Hip Abduction 15.3 P:Seated on the chair; E: Knee Extension 15.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes(parallel bar or back rest)

3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 16. Balance Training 16.1 P: Standing; E:Walk with Hip flexion 90o like soldier); S:No 16.2 P: Standing; E: Tandem Gait; S: Yes(parallel bar) 16.3 P: Standing; E: Step up and down; S: No 16.4 P: Seated on the chair; E:TUG habitual walk speed; S: No 16.5 P:Standing; E:Romberg- feet together; S: No+ ball reach

Strength Training 16.1 P: Ventral Decubitus; E: Hip Extension (Table position + raise one arm) 16.2 P:Lateral Decubitus; E: Hip Aduction 16.3 P:Standing; E: Squat; S:No 16.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest) 3 sets, 10 repetitions, 55-65% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

9a week

Day 17. Balance Training 17.1 P:Standing; E:Romberg- feet together; S: No+ ball reach 17.2 P: Standing; E: Step up and down; S: No 17.3 P: Seated on the chair; E:TUG habitual walk speed; S: No + Dual task (cognitive) 17.4 P: Standing; E:Walk (6 meters) increasing speed; S: No

Strength Training 17.1 P: Dorsal Decubitus; E:Hip Flexion 17.2 P:Lateral Decubitus; E: Hip Abduction 17.3 P:Seated on the chair; E: knee extension 17.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes (parallel bar or back rest) 3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 18. Balance Training 18.1 P:Standing; E:Romberg- feet together; S: No+ ball reach 18.2 P: Standing; E: Step up and down; S: No 18.3 P: Seated on the chair; E:TUG habitual walk speed; S: No + Dual task (cognitive) 18.4 P: Standing; E:Walk (6 meters) increasing step length; S: No

Strength Training 18.1 P: Ventral Decubitus; E: Hip Extension (Table position + raise arm and leg) 18.2 P:Lateral Decubitus; E: Hip Aduction 18.3 P:Standing; E: Split Squat; S:No; L:0.5 Kg 18.4 P: Standing; E: Knee Flexion; S: Yes (parallel bar or back rest)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

10a week

Day 19. Balance Training

19.1 P:Standing; E:Romberg- feet together; S: No+ Reach tasks 19.2 P: Standing E:Side step walking; S: No+ ball reach 19.3 P:Standing; E:Romberg- feet together; S: No+ unstable surface+ eyes opened and closed 19.4 P: Standing; E:Walk (6 meters) increasing step length; S: No Strength Training 19.1 P: Dorsal Decubitus; E:Hip Flexion 19.2 P:Lateral Decubitus; E: Hip Abduction 19.3 P:Seated on the chair; E: Knee Extension 19.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes (parallel bar or back res)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 20. Balance Training 20.1 P:Standing; E:Romberg- feet together; S: No+ Reach tasks 20.2 P: Standing; E:Side step walking; S: No+ ball reach 20.3 P: Standing; E: One leg stance; S: No + unstable surface 20.4 P: Standing; E:Walk (6 meters) with scapular dissociation and cervical rotation; S: No

Strength Training 20.1 P: Ventral Decubitus; E: Hip Extension (Table position + raise arm and leg) 20.2 P:Lateral Decubitus; E: Hip Aduction 20.3 P:Standing; E: Split Squat; S:No; L:0.5 Kg 20.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

11a week

Day 21. Balance Training

Circuit Training:

1. Stepping over barriers (Rolls, Steps)
2. Gait Training (increasing step length, changing speed, with scapular dissociation and cervical rotation)
3. Gait with motor tasks (Ball reach )
4. Balance Boards

Strength Training 21.1 P: Dorsal Decubitus; E:Hip Flexion 21.2 P:Lateral Decubitus; E: Hip Abduction 21.3 P:Seated on the chair; E: Knee Extension; S:Yes(parallel bar or back rest) 21.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes(parallel bar or back rest)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 22. Balance Training

Circuit Training:

1. Stepping over barriers (Rolls, Steps)
2. Gait Training (increasing step length, changing speed, with scapular dissociation and cervical rotation)
3. Gait with motor tasks (Ball reach)
4. Balance Boards

Strength Training

22.1 P: Ventral Decubitus; E: Hip Extension (Table position + raise arm and leg); L: 0.5 Kg 22.2 P:Lateral Decubitus 22.3 P:Standing; E: Split Squat; S:No; E: Hip Aduction; L:1.0 Kg 22.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

12a week

Day 23. Balance Training

Circuit Training:

1.1 Stepping over barriers (Rolls, Steps) 2.Gait Training (increasing step length, changing speed, with scapular dissociation and cervical rotation) 3.Gait with cognitive tasks 4.Balance Boards

Strength Training

23.1 P: Dorsal Decubitus; E:Hip Flexion 23.2 P:Lateral Decubitus; E: Hip Abduction 23.3 P:Seated on the chair; E: Knee Extension 23.4 P:Standing; E: Dorsiflexion/ Plantar Flexion; S:Yes (parallel bar or back rest)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

Day 24. Balance Training

Circuit Training:

1.1 Stepping over barriers (Rolls, Steps) 2.Gait Training (increasing step length, changing speed, with scapular dissociation and cervical rotation) 3.Gait with cognitive tasks 4.Balance Boards

Strength Training 24.1 P: Ventral Decubitus; E: Hip Extension (Table position + raise arm and leg); L: 0.5 Kg 24.2 P:Lateral Decubitus; E: Hip Aduction 24.3 P:Standing; E: Split Squat; S:No; L:0.5 Kg 24.4 P: Standing; E: Knee Flexion; S: Yes(parallel bar or back rest)

3 sets, 8 repetitions, 65-75% RM

P: Position ; E: Exercise ; S: Support; A: Accessory; L: Load ; RM: Repetition Maximum

ELIGIBILITY:
Inclusion Criteria:

* volunteers above the age of 65 who are community residents and classified as frail according to the criteria established by Fried et al. will be selected for inclusion in the study

Exclusion Criteria:

* previous lower extremities orthopedic surgery, a history of fractures within the past year, an inability to walk unaided, carriers of neurological diseases, diagnosed acute inflammatory disease that could interfere in the assessments and the program, tumor growth in the last five years and cognitive impairment based on the mini-mental state examination [4]. Moreover, will be excluded volunteers who are absent more than three consecutive training and / or more than 25% of the sessions, and / or present the course of the physical program changes or decompensation and / or disease injury.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
strength muscle evaluation | baseline
  The Elbow flexors and extensors, trunk flexors and extensors, hip abductor and adductor, knee flexors and extensors and ankle dorsiflexors and plantarflexors muscle strength of the dominant limb will be evaluated by an isokinetic dynamometer
Balance | baseline
  Balance in semi-static stance was measured using the force platform. Data on 6 stances were collected for each subject: standing on a fixed platform with eyes open and closed; standing on an unstable platform with eyes open and closed; and in single-leg stance with eyes open on the right leg and on the left leg.
gait | baseline
  The gait parameters will be analyzed using the GAITRite Platinum 26' Portable Walkway System to evaluated spatial and temporal gait variables.
functional performance | baseline
  Timed Up and Go (TUG) test will be used.

SECONDARY OUTCOMES:
strength muscle evaluation | change from baseline in 3 months
  The Elbow flexors and extensors, trunk flexors and extensors, hip abductor and adductor, knee flexors and extensors and ankle dorsiflexors and plantarflexors muscle strength of the dominant limb will be evaluated by an isokinetic dynamometer
Balance | change from baseline in 3 months
  Balance in semi-static stance was measured using the force platform. Data on 6 stances were collected for each subject: standing on a fixed platform with eyes open and closed; standing on an unstable platform with eyes open and closed; and in single-leg stance with eyes open on the right leg and on the left leg.
gait | change from baseline in 3 months
  The gait parameters will be analyzed using the GAITRite Platinum 26' Portable Walkway System to evaluated spatial and temporal gait variables.
functional performance | change from baseline in 3 months
  Timed Up and Go (TUG) test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela CC de Abreu, Professor, Study Chair — School of Medicine of RibeirãoPreto, University of São Paulo, FMRP-USP

IPD SHARING:
Plan to Share IPD: Yes
After the end of the protocol and the data evaluation, the results will be send to each participant.

REFERENCES:
- [Background] de Labra C, Guimaraes-Pinheiro C, Maseda A, Lorenzo T, Millan-Calenti JC. Effects of physical exercise interventions in frail older adults: a systematic review of randomized controlled trials. BMC Geriatr. 2015 Dec 2;15:154. doi: 10.1186/s12877-015-0155-4. PMID 26626157
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Lustosa LP, Coelho FM, Silva JP, Pereira DS, Parentoni AN, Dias JM, Dias RC, Pereira LS. The effects of a muscle resistance program on the functional capacity, knee extensor muscle strength and plasma levels of IL-6 and TNF-alpha in pre-frail elderly women: a randomized crossover clinical trial--a study protocol. Trials. 2010 Jul 28;11:82. doi: 10.1186/1745-6215-11-82. PMID 20667082
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Ashfield TA, Syddall HE, Martin HJ, Dennison EM, Cooper C, Aihie Sayer A. Grip strength and cardiovascular drug use in older people: findings from the Hertfordshire Cohort Study. Age Ageing. 2010 Mar;39(2):185-91. doi: 10.1093/ageing/afp203. Epub 2009 Dec 17. PMID 20019032
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] McPhee JS, French DP, Jackson D, Nazroo J, Pendleton N, Degens H. Physical activity in older age: perspectives for healthy ageing and frailty. Biogerontology. 2016 Jun;17(3):567-80. doi: 10.1007/s10522-016-9641-0. Epub 2016 Mar 2. PMID 26936444
- [Background] Gobbens RJ, Luijkx KG, Wijnen-Sponselee MT, Schols JM. Toward a conceptual definition of frail community dwelling older people. Nurs Outlook. 2010 Mar-Apr;58(2):76-86. doi: 10.1016/j.outlook.2009.09.005. PMID 20362776
- [Background] Gine-Garriga M, Guerra M, Pages E, Manini TM, Jimenez R, Unnithan VB. The effect of functional circuit training on physical frailty in frail older adults: a randomized controlled trial. J Aging Phys Act. 2010 Oct;18(4):401-24. doi: 10.1123/japa.18.4.401. PMID 20956842
- [Background] Gine-Garriga M, Guerra M, Unnithan VB. The effect of functional circuit training on self-reported fear of falling and health status in a group of physically frail older individuals: a randomized controlled trial. Aging Clin Exp Res. 2013 Jun;25(3):329-36. doi: 10.1007/s40520-013-0048-3. Epub 2013 May 17. PMID 23740589
- [Background] Aguirre LE, Villareal DT. Physical Exercise as Therapy for Frailty. Nestle Nutr Inst Workshop Ser. 2015;83:83-92. doi: 10.1159/000382065. Epub 2015 Nov 2. PMID 26524568
- [Background] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Fairhall N, Sherrington C, Lord SR, Kurrle SE, Langron C, Lockwood K, Monaghan N, Aggar C, Cameron ID. Effect of a multifactorial, interdisciplinary intervention on risk factors for falls and fall rate in frail older people: a randomised controlled trial. Age Ageing. 2014 Sep;43(5):616-22. doi: 10.1093/ageing/aft204. Epub 2013 Dec 30. PMID 24381025
- [Background] Lustosa LP, Silva JP, Coelho FM, Pereira DS, Parentoni AN, Pereira LS. Impact of resistance exercise program on functional capacity and muscular strength of knee extensor in pre-frail community-dwelling older women: a randomized crossover trial. Rev Bras Fisioter. 2011 Aug-Sep;15(4):318-24. English, Portuguese. PMID 21971726
- [Background] Cadore EL, Casas-Herrero A, Zambom-Ferraresi F, Idoate F, Millor N, Gomez M, Rodriguez-Manas L, Izquierdo M. Multicomponent exercises including muscle power training enhance muscle mass, power output, and functional outcomes in institutionalized frail nonagenarians. Age (Dordr). 2014 Apr;36(2):773-85. doi: 10.1007/s11357-013-9586-z. Epub 2013 Sep 13. PMID 24030238
- [Background] Kim H, Suzuki T, Kim M, Kojima N, Ota N, Shimotoyodome A, Hase T, Hosoi E, Yoshida H. Effects of exercise and milk fat globule membrane (MFGM) supplementation on body composition, physical function, and hematological parameters in community-dwelling frail Japanese women: a randomized double blind, placebo-controlled, follow-up trial. PLoS One. 2015 Feb 6;10(2):e0116256. doi: 10.1371/journal.pone.0116256. eCollection 2015. PMID 25659147
- [Background] 20. Porto JM, Marques NR, Junior RCF, de Abreu DCC: The effect of foot support on trunk strength assessment using isokinetic dynamometry. Isok and Exerc Scien. 2015;23:283-289.
- [Background] Gomes MM, Reis JG, Carvalho RL, Tanaka EH, Hyppolito MA, Abreu DC. Analysis of postural control and muscular performance in young and elderly women in different age groups. Braz J Phys Ther. 2015 Jan-Feb;19(1):1-9. doi: 10.1590/bjpt-rbf.2014.0068. Epub 2015 Feb 3. PMID 25651132
- [Background] Tanaka EH, Santos PF, Reis JG, Rodrigues NC, Moraes R, Abreu DC. Is there a relationship between complaints of impaired balance and postural control disorder in community-dwelling elderly women? A cross-sectional study with the use of posturography. Braz J Phys Ther. 2015 May-Jun;19(3):186-93. doi: 10.1590/bjpt-rbf.2014.0086. Epub 2015 Jun 12. PMID 26083602
- [Background] Freire Junior RC, Porto JM, Rodrigues NC, Brunelli RM, Braga LF, de Abreu DC. Spatial and temporal gait characteristics in pre-frail community-dwelling older adults. Geriatr Gerontol Int. 2016 Oct;16(10):1102-1108. doi: 10.1111/ggi.12594. Epub 2015 Sep 3. PMID 26338502
- [Background] 24. Kochi MN, Marques NR, da Costa GC, Reis JG, de Paula FJA, Ferreira CHJ, de Abreu DCC: Impact of First 10 Years of Post Menopause on Muscle Function, Muscle Mass and Bone Mineral Density in Adult Women. J Osteopor Phys Act. 2015;3:3.
- [Background] Santos ML, Gomes WF, Pereira DS, Oliveira DM, Dias JM, Ferrioli E, Pereira LS. Muscle strength, muscle balance, physical function and plasma interleukin-6 (IL-6) levels in elderly women with knee osteoarthritis (OA). Arch Gerontol Geriatr. 2011 May-Jun;52(3):322-6. doi: 10.1016/j.archger.2010.05.009. PMID 20627334
- [Background] Chen TC, Chen HL, Lin MJ, Wu CJ, Nosaka K. Muscle damage responses of the elbow flexors to four maximal eccentric exercise bouts performed every 4 weeks. Eur J Appl Physiol. 2009 May;106(2):267-75. doi: 10.1007/s00421-009-1016-7. Epub 2009 Mar 5. PMID 19263073
- [Background] 28. Antero-Jacquemin JS, Santos P, Garcia PA, Dias RC, Dias JMD: Comparacao da funcao muscular isocinética dos membros inferiores entre idosos caidores e não caidores. Fisioter Pesq. 2012;19:39-44.
- See also: World Health Organization. Active ageing: a policy framework. — http://apps.who.int/iris/bitstream/10665/67215/1/WHO_NMH_NPH_02.8.pdf